CLINICAL TRIAL: NCT04854928
Title: A Double-blind, Placebo-controlled, Interventional Parallel Group Study to Evaluate the Antiviral Effect of a Single Nasal Application of LTX-109 3% Gel, in Comparison to Placebo Gel, in Subjects With COVID-19 Infection.
Brief Title: Study to Evaluate a Single Dose of LTX-109 in Subjects With COVID-19 (Coronavirus Disease 2019) Infection.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharma Holdings AS (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C21-109-09
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: LTX-109; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomised, Double-blind, Placebo-controlled Randomization 1:1, active to placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTX-109 treatment (Experimental): Single Dose by Nasal application of LTX-109 gel 3%, 250 microliters in each nostril.
  Interventions: Drug: LTX-109 gel, 3%
- Placebo (Placebo Comparator): Single Dose by Nasal application of placebo gel, 250 microliters in each nostril.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: LTX-109 gel, 3% — A Single dose of LTX-109 gel will be applied topically to both nostrils by a qualified health professional. A large drop of IMP will be applied into each nostril and distributed to cover the whole area of the nostril.
  Arms: LTX-109 treatment
Drug: Placebo gel — A Single dose of placebo gel will be applied topically to both nostrils by a qualified health professional. A large drop of IMP will be applied into each nostril and distributed to cover the whole area of the nostril.
  Arms: Placebo

SUMMARY:
A Phase IIa, double-blind, placebo-controlled, randomised study designed to evaluate the effect, safety and tolerability of LTX-109 administered topically to the anterior nares in subjects with COVID-19 infection.

DETAILED DESCRIPTION:
A total of 60 subjects will be randomised to achieve approximately 46 completed and evaluable subjects. Subjects will be randomised 1:1 to one single dose of either active treatment or placebo.

All potential study subjects will be contacted and invited to a screening video-call with the Investigator. Full verbal information will be given and the consent for participation in the study will be signed electronically.

Eligible subjects will be visited twice at home by a study nurse on Day 1. During the first visit, one standard deep nose swab (one nostril) and one from the anterior part of the nose (both nostrils) will be collected. Symptom score will be assessed by the subject before dosing. The investigational medicinal product (IMP) will then be applied topically to both nostrils by the study nurse.

The study nurse will come back to collect nasal swab samples 2 hours after administration of the IMP, using the same sampling procedure as for the baseline samples.

Subjects will use an electronic diary for daily registrations of adverse events, concomitant medications and symptom score until Day 7.

A follow-up phone contact will be performed 7 days after IMP administration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give electronically signed informed consent for participation in the study.
2. Male or female subject ≥18 years of age at screening.
3. Women of child-bearing potential have to agree to use an acceptable birth control method during participation in the investigation and a negative pregnancy test (beta human chorionic gonadotropin dipstick test in urine) at Day 1 will be required.
4. A positive PCR test (polymerase chain reaction test) or antigen test for SARS-CoV-2. The positive result must be available no later than 4 days from initiation of symptoms, if any.
5. Duration of symptoms not exceeding 6 days prior to baseline/IMP administration (Day 1).
6. Access to a mobile phone or computer and ability to use the electronic diary application and to participate in web-based appointments.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Other upper respiratory tract infection with concomitant symptoms that can influence the results, such as sinusitis or tonsillitis.
3. Known allergy or hypersensitivity to the components of the IMP.
4. Current use of immunosuppressive therapy within the last 4 weeks prior to Day 1 and during the study.
5. Current use of nasally administered drugs within the last 2 weeks prior to Day 1 and during the study.
6. Vaccinated against COVID-19 or scheduled for vaccination within the study period.
7. Previous COVID-19 infection.
8. Any systemic anti-viral treatment within the last 4 weeks prior to Day 1 and during the study.
9. Pregnant, nursing or actively trying to conceive a child.
10. Inability to take medications nasally.
11. In situ nasal jewellery or open nasal piercings.
12. Planned treatment or treatment with another investigational drug within 30 days prior to Day 1. Subjects consented and screened but not dosed in previous Phase I studies are not excluded.
13. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2 ) viral load in the deep nasal cavity as measured by the amount of live virus in the samples. | From baseline (pre-dose) to 2 hours (h) post-dose
  Assessment of viral load at baseline (pre-dose) and 2h post-dose to evaluate the effect of a single dose of LTX-109 nasal gel as compared to placebo. Reduction in SARS-CoV-2 viral load is measured by a standardised reverse transcription quantitative polymerase chain reaction (RT-qPCR) method and virus titration followed by cell viability assay to quantify the amount of live virus in the samples (Median Tissue Culture Infectious Dose [TCID50]). Viral load will be expressed as TCID50/mL.

SECONDARY OUTCOMES:
Reduction in SARS-CoV-2 viral load in the anterior nasal cavity as measured by the amount of live virus in the samples. | From baseline (pre-dose) to 2 hours (h) post-dose
  Assessment of viral load at baseline (pre-dose) and 2h post-dose to evaluate the effect of a single dose of LTX-109 nasal gel as compared to placebo. Reduction in SARS-CoV-2 viral load is measured by a standardised RT-qPCR method and virus titration followed by cell viability assay to quantify the amount of live virus in the samples, TCID50. Viral load will be expressed as TCID50/mL.
Assessment of safety and tolerability by frequency and seriousness of Adverse Events (AE) | From dosing until 7 days after dose.
  The Investigator will assess the seriousness of all AE according to the common definition of Serious Adverse Events (SAE). Frequency of AEs and SAEs will be summarised by treatment and overall.
Assessment of safety and tolerability by intensity of AE | From dosing until 7 days after dose.
  The Investigator will assess the intensity of an AE on a 5 graded scale. Grade refers to the severity of the AE, from Grade 1 (mild) through Grade 5 (death).

OTHER OUTCOMES:
Change in Symptom score for frequency of COVID-19 infection symptoms. | From pre-dose on Day 1 until Day 7.
  Daily assessments of frequency of symptoms using a study-specific questionnaire with 10 questions/symptoms. Symptoms included are fever, cough, trouble breathing, loss of smell or taste, nasal congestion or runny nose, sore throat and/or difficulty swallowing, headache, muscle and/or joint pain, stomach-ache and/or nausea and diarrhoea. The frequency of each symptom will be graded by the Subject using a 5 graded scale from Grade 1 (None of the time) through Grade 5 (All of the time). For each symptom, the absolute and percent change from baseline to Day 7 will be calculated.
Change in Symptom score for intensity of COVID-19 infection symptoms. | From pre-dose on Day 1 until Day 7.
  Daily assessments of intensity of symptoms using a study-specific questionnaire with 10 questions/symptoms. Symptoms included are fever, cough, trouble breathing, loss of smell or taste, nasal congestion or runny nose, sore throat and/or difficulty swallowing, headache, muscle and/or joint pain, stomach-ache and/or nausea and diarrhoea. The intensity of each symptom will be graded by the Subject using a 5 graded scale from Grade 1 (Not at all intense) through Grade 5 (Terribly intense). For each symptom, the absolute and percent change from baseline to Day 7 will be calculated.
Reduction in SARS-CoV-2 viral load in the deep nasal cavity as measured by qPCR. | From baseline (pre-dose) to 2 hours (h) post-dose
  Assessment of viral load at baseline (pre-dose) and 2h post-dose to evaluate the effect of a single dose of LTX-109 nasal gel as compared to placebo. Reduction in SARS-CoV-2 viral load is measured by a qPCR. Viral load will be expressed as log10 RNA copies per 1000 cells.
Reduction in SARS-CoV-2 viral load in the anterior nasal cavity as measured by qPCR. | From baseline (pre-dose) to 2 hours (h) post-dose
  Assessment of viral load at baseline (pre-dose) and 2h post-dose to evaluate the effect of a single dose of LTX-109 nasal gel as compared to placebo. Reduction in SARS-CoV-2 viral load is measured by a qPCR. Viral load will be expressed as log10 RNA copies per 1000 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lütken, MD, Study Director — Pharma Holdings AS
Locations (1):
- ClinSmart Sweden AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No